CLINICAL TRIAL: NCT04033549
Title: Utility of Thoracic Ultrasound in Patients With Acute Pancreatitis as a Prognostic Tool of Respiratory Dysfunction and Severity
Brief Title: Thoracic Ultrasound on Acute Pancreatitis
Acronym: ECOPANC
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. med. Hector Eloy Tamez Perez, Clinical Professor, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: GA18-00005
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Acute Pancreatitis
Keywords: Acute pancreatitis; Thoracic ultrasound
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Authors design a prospective, longitudinal, descriptive study to identify the findings of thoracic point-of-care ultrasound in patients with acute pancreatitis. Patients will be included in the study since August through December 2019, admitted to the University Hospital, "Dr. José E. González", Universidad Autonoma de Nuevo León. These patients will undergo a pulmonary and vena cava ultrasound at admission, at 24 and 48 hours. The authors will describe findings of pulmonary ultrasound and their correlation with severity in patients with acute pancreatitis of all etiologies. The authors will analyze variables such Systemic inflammatory response syndrome, severity according to the revised Atlanta criteria (2012), and systemic complications.

DETAILED DESCRIPTION:
Acute pancreatitis has been described as the most common cause of pancreatic disease with a global incidence of 33-74 per 100.000 people and a mortality of 1-16 per 100.000. Hydration with the purpose of preventing hypovolemia and hypoperfusion of organs is the cornerstone of initial disease management. "Aggressive" hydration, has been based on animal models and observational data from clinical studies, and has been associated with respiratory complications, compartment syndrome, sepsis, and mortality. Nowadays pulmonary ultrasound has been used in a wide array of clinical settings such as intensive care unit, emergency medicine, and nephrology. It has been a standardized tool in internal and pulmonary medicine.

Authors design a prospective, longitudinal, descriptive study to identify the findings of thoracic point-of-care ultrasound in patients with acute pancreatitis. Patients will be included in the study since August through December 2019, admitted to the University Hospital, "Dr. José E. González", Universidad Autonoma de Nuevo León.

OBJECTIVES

1. Primary objective:

   Describe findings of pulmonary ultrasound and their correlation with severity in patients with acute pancreatitis of all etiologies. The authors will analyze variables such Systemic inflammatory response syndrome, severity according to the revised Atlanta criteria (2012), and systemic complications.
2. Secondary objectives:

   1. to correlate the number of B-type lines measured by thoracic point-of-care ultrasound with severity in patients with acute pancreatitis.
   2. to correlate the diameter in centimeters of inferior vena cava measured by thoracic point-of-care ultrasound with severity in patients with acute pancreatitis
   3. to correlate the inferior vena cava diameter with the 48 hours post-admission mortality rate in patients with acute pancreatitis.

STUDY DESIGN Prospective, transversal, descriptive.

SUBJECTS AND METHODS

1. Patients:

   In the time period of August 2019 through December 2019 the authors will include patients with pancreatitis.

   The investigators will include all patients that attend the Emergency department of Hospital Universitario, "Dr. José Eleuterio González" U.A.N.L, with a diagnosis of acute pancreatitis of all causes.

   Inclusion criteria:
   1. Patients with diagnosis of acute pancreatitis by means of clinical presentation, laboratory results and/or imaging.
   2. Both genders.
   3. All etiologies of pancreatitis.
   4. Ages above 18.

   Exclusion criteria:
   1. History of acute pancreatitis in prior 12 months.
   2. Patients with referrals from other institutions.
   3. Patients with other chronic comorbidities such as renal or cardiac insufficiency.
   4. Patients with acute pancreatitis and high suspicion of cholangitis.
   5. Patients with acute pancreatitis and acute cholecystitis.
   6. Pregnant patients with acute pancreatitis.
   7. Patients who decline being part of this study.
2. Methods:

The investigators will study all patients who come to the emergency room of the hospital with diagnosis of Acute Pancreatitis. Patients will undergo a pulmonary and vena cava ultrasound at admission, at 24 and 48 hours.

Ultrasound will be performed bilateral intercostal with the patient in supine decubitus with the head at 30 degrees, after the application of acoustic gel on the skin. To improve imaging, the intercostal spaces will be extended by raising the ipsilateral arm of each patient to the level of the head or above it during the procedure.

Each hemithorax is divided into 4 areas: anterior and lateral, superior and inferior. For each hemithorax, the anterior area was delineated between the clavicle and the diaphragm and from the parasternal line to the anterior axillary line. The lateral area was delineated between the axilla and the diaphragm and from the anterior to the posterior axillary line. The upper quadrants were demarcated from the 1st to the 3rd intercostal space and the lower quadrants from the 4th to the 6th intercostal space. A total of 8 areas of the chest will be visualized during normal breathing.

Findings that will be reported upon pulmonary ultrasound:

B lines: They are hydro-aerial artifacts in comet tail image, begin at the pleural line, are hyperechoic, well defined, disseminated towards the end of the screen, delete A lines , and accompany pleural movements.

The lines separated from each other around 7 mm correspond to interstitial edema, while those that distance 3 mm indicate the presence of alveolar edema. The presence of more than 3 B lines indicate the presence of an alveolar-interstitial syndrome.

Pleural effusion: It is visualized as a space free of echoes (anechoic image, "black") between the visceral pleura (pulmonary line), together with the parietal pleura (pleural line) and the shadow of the ribs. In M mode, the movement of the lung line or the visceral pleura to the pleural line or the parietal pleura upon inspiration is shown, creating the sinusoidal sign.

Measurement of the inferior Vena cava:

Intravascular volume status will be assessed by measuring the diameter and percentage of collapse of the inferior vena cava. It is performed in the subxiphoid window with the identification of the four cardiac chambers, then a 90º turn of the transducer is made in the cephalad direction, which shows the right atrium, the mouth of the vena cava and the hepatic gland above it. To measure its diameter, it will be beyond the confluence point of the hepatic veins, which is usually found approximately 2 cm from the mouth of the inferior vena cava-right atrium. Based on the measurement and collapse of the IVC, volemic state will be defined in a patient with spontaneous breathing as follows: a diameter of the Inferior cava vein <2 cm that collapses> 50% suggests lack of volume; however, a diameter of the Inferior cava vein > 2 cm that collapses <50% suggests a hypervolemic state.

The authors will analyze variables such Systemic inflammatory response syndrome, severity according to the revised Atlanta criteria (2012), and systemic complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of acute pancreatitis by means of clinical presentation, laboratory results and/or imaging.
* Both genders.
* All etiologies of pancreatitis.
* Ages above 18.

Exclusion Criteria:

* History of acute pancreatitis in prior 12 months.
* Patients with referrals from other institutions.
* Patients with other chronic comorbidities such as renal or cardiac insufficiency.
* Patients with acute pancreatitis and high suspicion of cholangitis.
* Patients with acute pancreatitis and acute cholecystitis.
* Pregnant patients with acute pancreatitis.
* Patients who decline being part of this study.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients that attend the Emergency department of Hospital Universitario, "Dr. José Eleuterio González" U.A.N.L, with a diagnosis of acute pancreatitis of all causes
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
B-type lines on thoracic point-of-care ultrasound in patients with acute pancreatitis | 48 hours
  The number of B-type lines measured by thoracic point-of-care ultrasound in patients with acute pancreatitis.

SECONDARY OUTCOMES:
Diameter of inferior vena cava on thoracic point-of-care ultrasound in patients with acute pancreatitis. | 48 hours
  The diameter in centimeters of inferior vena cava measured by thoracic point-of-care ultrasound in patients with acute pancreatitis
B-type lines and Atlanta score in patients with acute pancreatitis | 48 hours
  To correlate the presence of B-type lines on thoracic point-of-care ultrasound with Atlanta score in patients with acute pancreatitis
Inferior vena cava diameter and Atlanta score in patients with acute pancreatitis | 48 hours
  To correlate the inferior vena cava diameter with the Atlanta score in patients with acute pancreatitis
Inferior vena cava diameter and 48 hours mortality in patients with acute pancreatitis | 7 days
  To correlate the inferior vena cava diameter with the 48 hours post-admission mortality rate in patients with acute pancreatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Cuellar Monterrubio, M.D., Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Hospital Universitario Dr. Jose E. Gonzalez, Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes
If need information will be available upon email contact request.
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: email contact request for academic purposes